CLINICAL TRIAL: NCT02685722
Title: Umbilical Cord Mesenchymal Stem Cells Between Gel Treatment Difficult Skin Ulcer Healing Efficacy and Safety of Random, Open, Before-and-after Study
Brief Title: UC-MSCs Gel Treatment Difficult Healing of Skin Ulcers
Acronym: UC-MSCs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-ST-008
Record Dates: First submitted 2016-01-21; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Difficult to Healing of Skin Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UC-MSCs Gel group (Experimental): This study for a six-month trials,Randomized, open, and parallel comparison before and after its own,Stage test includes screening stage, stochastic screening of more than a month difficult to heal wounds 20 people.treatment period and follow-up period.In accordance with chronic wound criteria for the patient,By producing the principle of random number,Were randomly divided into UC-MSCs Gel group or Gel group,The researchers according to the situation of wound healing time and decided to use the secondary treatment,to observe the clinical efficacy and safety.
  Interventions: Biological: UC-MSCs Gel group
- Gel group (Experimental): This study for a six-month trials,Randomized, open, and parallel comparison before and after its own,Stage test includes screening stage, stochastic screening of more than a month difficult to heal wounds 20 people.treatment period and follow-up period.In accordance with chronic wound criteria for the patient,By producing the principle of random number,Were randomly divided into UC-MSCs Gel group or Gel group,The researchers according to the situation of wound healing time and decided to use the secondary treatment,to observe the clinical efficacy and safety.
  Interventions: Other: Gel group

INTERVENTIONS:
Biological: UC-MSCs Gel group — This study for a six-month trials,Randomized, open, and parallel comparison before and after its own,Stage test includes screening stage, stochastic screening of more than a month difficult to heal wounds 20 people.By generating a random number of principle,Observation of UC-MSCs Gel group patients efficacy, safety and tolerability of selective parameter.
  Arms: UC-MSCs Gel group
Other: Gel group — This study for a six-month trials,Randomized, open, and parallel comparison before and after its own,Stage test includes screening stage, stochastic screening of more than a month difficult to heal wounds 20 people.By generating a random number of principle,observed and compared Gel group patients may be no efficacy.
  Arms: Gel group

SUMMARY:
This study for a six-month trials, Randomized, open, and parallel comparison before and after its own, Stage test includes screening stage, treatment period and follow-up period. In accordance with chronic wound criteria for the patient, By producing the principle of random number, Were randomly divided into UC-MSCs Gel group or Gel group, The researchers according to the situation of wound healing time and decided to use the secondary treatment, To observe the clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 year old male or female (pregnancy);
* Has the ability to care for, has the ability to self signed informed consent, 7 to 17 years of age must be signed by the guardian informed consent;
* The process of psychological stability, can finish the tes

Exclusion Criteria:

* Allergic constitution, or known allergic to pork or beef source products, gao min physique person;
* The wound is more than 10 cm by 10 cm;
* People with mental illness, drug abusers and or other items;
* 1 month used or are using the sugar metabolism of drugs, such as corticosteroids, thiazide diuretics, tricyclic antidepressants, etc;
* 3 month participated in other similar test;
* Serious infectious disease not controller;
* With surgery, such as severe trauma stress situation;
* Always had a history of tumor;
* Clinical researchers or for other reasons can't cooperate with the doctors, and other information is not suitable for clinical study of patients.

Ages: 17 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 6 months
  Frequency and severity of Adverse Events

SECONDARY OUTCOMES:
Relative Wound Area Regression of 40% or More at 6 Week | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: xiaobing Fu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China